CLINICAL TRIAL: NCT05281562
Title: Effects of Supplemental Immunonutrition on Healing of Chronic Non-Healing Lower Extremity Ulcers in Diabetic Patients: A Pilot Study
Brief Title: Immunonutrition for Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Not enough patients meeting eligibility criteria to complete the study. It took months from study initiation to enroll 1 participant in February 2023. Once it was clear it was not possible to enroll another participant, the study was terminated.
Sponsor: Prisma Health-Midlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1876718
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus; Diabetic Peripheral Neuropathy; Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot | interventions — Omacor; Fatty Acids, Omega-3; Arginine; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive 6 weeks of oral immunonutrition supplementation, consisting of L-Arginine, Vitamin C, and Omega-3 fatty acids, in addition to standard of care for wound treatment or standard of care alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care Group (No Intervention): Patients will receive standard of care wound treatment as determined by a treating physician.
- Immunonutrition Supplementation Group (Experimental): Patients will receive a 6 week daily oral supply of 1.68 grams Omega-3 fatty acids, 4.5 grams L-Arginine, and 500 mg Vitamin C.
  Interventions: Drug: Lovaza; Drug: L-Arginine Powder; Drug: Vitamin C

INTERVENTIONS:
Drug: Lovaza — Daily dose of 1.68grams omega-3 fatty acids, 2 Lovaza pills per day.
  Other Names: omega-3 fatty acids; omega-3-acid ethyl esters
  Arms: Immunonutrition Supplementation Group
Drug: L-Arginine Powder — Daily dose of 4.5 grams L-Arginine, powder form.
  Other Names: Arginine; 2-amino-5-guanidinopentanoic acid
  Arms: Immunonutrition Supplementation Group
Drug: Vitamin C — Daily dose of 500 mg Vitamin C, powder form.
  Other Names: Ascorbic acid
  Arms: Immunonutrition Supplementation Group

SUMMARY:
Diabetes-induced peripheral neuropathy can lead to the development of diabetic foot ulcers (DFUs), which can have a devastating effect on patients' lives and can lead to life threatening infection, amputations, and even death. Conventional treatment of DFUs are time consuming, burdensome, costly, and often do not treat the root cause of the problem. Even with proper care, ulcers can take a significantly longer time to heal in diabetic patients due to the altered physiology which does not allow for the proper nutrients and healing factors to mobilize to the site of injury, leaving these ulcers with a poor chance of healing and at high risk for infection and possible amputation. Supplemental immunonutrition therapy may offer a viable, low cost, rapidly scalable, and widely available approach to enhance the body's ability to heal itself. This prospective, randomized pilot study will evaluate the effect of a 6-week daily oral course of a specific combination of immunonutrients, L-Arginine, Omega-3 fatty acids, and Vitamin C, on wound healing in diabetic patients with chronic lower extremity ulcers compared to traditional standard of care. The deliverables of this clinical project will serve to advance a cost-effective added strategy to address a significant unmet clinical need in treatment for the diabetic patient population. Study outcomes will lay the foundation for a multi-site clinical trial to establish the efficacy and cost-effectiveness of this strategy across the health care system.

DETAILED DESCRIPTION:
Diabetes mellitus is one of the most prevalent chronic diseases in the world and its incidence is expected to increase over the next 20 years. Historically there are three described types of diabetes mellitus: Type 1, Type 2, and Gestational. The etiology of disease may vary between types, and our current understanding notes overlap of these types, yet the resulting pathophysiology is the same: poor peripheral blood flow, decreased cellular response at the injury site, elevated glucose levels, and poor nutrient transport. Despite many of these patients having an elevated Body Mass Index (BMI), they are functionally under or malnourished. In addition, some patients develop progressive neurologic dysfunction, called peripheral neuropathy (PN). A common complication of diabetes induced PN is the development of diabetic foot ulcers (DFUs), which can have a devastating effect on patients' lives and can lead to life threatening infection, amputations, and even death.

Conventional treatment of DFUs includes shoe wear modification, self-monitoring, local wound care, brace and shoe offloading, and surgical intervention as well as more sophisticated treatments such as bioengineered cellular technologies and hyperbaric oxygen therapy. These modalities are time consuming, burdensome, costly, and often do not treat the root cause of the problem. Additionally, even with proper care, ulcers can take a significantly longer time to heal in diabetic patients due to the altered physiology which does not allow for the proper nutrients and healing factors to mobilize to the site of injury, leaving these ulcers with a poor chance of healing and at high risk for infection and possible amputation. In contrast to traditional treatment modalities, nutrition therapy has been shown to aide in healing of chronic wounds by providing essential nutrients which were not previously present in necessary amounts in diabetic patients. Nutrition therapy has proven useful in modulating inflammation and the immune response, optimizing glucose control, and attenuating the hypermetabolic response to ulcers, ultimately improving healing and recovery. Thus, supplemental immunonutrition therapy may offer a viable, low cost, rapidly scalable, and widely available approach to enhance the body's ability to heal itself.

This prospective, randomized pilot study will evaluate the effect of a 6-week daily oral course of a specific combination of immunonutrients, L-Arginine, Omega-3 fatty acids, and Vitamin C, on wound healing in diabetic patients with chronic lower extremity ulcers compared to traditional standard of care. Wound characteristics and clinical photographs will be documented throughout the course of the study. Patient-reported pain scores, side effects, and unscheduled visits to emergency departments/urgent care centers will be recorded. Patients randomized to receive immunonutrition supplementation will complete an additional survey detailing their satisfaction with the treatment plan upon completion of their participation in the study. The deliverables of this clinical project will serve to advance a cost-effective added strategy to address a significant unmet clinical need in treatment for the diabetic patient population. Study outcomes will lay the foundation for a multi-site clinical trial to establish the efficacy and cost-effectiveness of this strategy across the health care system.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of informed consent
* Toe blood pressure (TBP) >40 mmHg
* Hemoglobin A1c <10% (measured within the previous 6 months)
* Diagnosis of diabetes mellitus
* Presence of at least one new chronic, non-healing (present for ≥4 weeks), lower extremity wound (Werner stage 2-3)
* Documented lipid panel within 3 months of study enrollment
* Documented CMP within 3 months of study enrollment
* Documented ECG within 3 months of study enrollment
* Receiving standard or care defined as sharps debridement, appropriate dressing, and offloading.

Exclusion Criteria:

* Allergy to fish
* Current smoker
* Currently taking any OTC supplements containing Omega-3 fatty acids, L-Arginine, or Vitamin C, or antibiotics
* Presence of at least one of the following diseases or conditions: End stage renal disease as defined by patients who have been diagnosed with Stage 4 kidney disease and are not on hemodialysis or who are on hemodialysis with a GFR consistently < 15L/min and BUN > 60, Untreated deep bone infection (osteomyelitis), Currently pregnant or breastfeeding
* Women of child-bearing potential
* Prisoners and other institutionalized individuals
* Any patients who have a legal representative to make medical decisions on their behalf or any individuals who are otherwise deemed as medically incompetent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Benjamin Jackson, MD, Principal Investigator — Prisma Health-Midlands
Locations (1):
- Prisma Health, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deshpande AD, Harris-Hayes M, Schootman M. Epidemiology of diabetes and diabetes-related complications. Phys Ther. 2008 Nov;88(11):1254-64. doi: 10.2522/ptj.20080020. Epub 2008 Sep 18. PMID 18801858
- [Background] Allen L, Powell-Cope G, Mbah A, Bulat T, Njoh E. A Retrospective Review of Adverse Events Related to Diabetic Foot Ulcers. Ostomy Wound Manage. 2017 Jun;63(6):30-33. PMID 28657897
- [Background] Corriere M, Rooparinesingh N, Kalyani RR. Epidemiology of diabetes and diabetes complications in the elderly: an emerging public health burden. Curr Diab Rep. 2013 Dec;13(6):805-13. doi: 10.1007/s11892-013-0425-5. PMID 24018732
- [Background] Hicks CW, Selvin E. Epidemiology of Peripheral Neuropathy and Lower Extremity Disease in Diabetes. Curr Diab Rep. 2019 Aug 27;19(10):86. doi: 10.1007/s11892-019-1212-8. PMID 31456118
- [Background] Rice JB, Desai U, Cummings AK, Birnbaum HG, Skornicki M, Parsons NB. Burden of diabetic foot ulcers for medicare and private insurers. Diabetes Care. 2014;37(3):651-8. doi: 10.2337/dc13-2176. Epub 2013 Nov 1. PMID 24186882
- [Background] Evans DC, Martindale RG, Kiraly LN, Jones CM. Nutrition optimization prior to surgery. Nutr Clin Pract. 2014 Feb;29(1):10-21. doi: 10.1177/0884533613517006. Epub 2013 Dec 17. PMID 24347529
- [Background] Alexander JW, Supp DM. Role of Arginine and Omega-3 Fatty Acids in Wound Healing and Infection. Adv Wound Care (New Rochelle). 2014 Nov 1;3(11):682-690. doi: 10.1089/wound.2013.0469. PMID 25371851
- [Background] Zhang XJ, Chinkes DL, Wolfe RR. The anabolic effect of arginine on proteins in skin wound and muscle is independent of nitric oxide production. Clin Nutr. 2008 Aug;27(4):649-56. doi: 10.1016/j.clnu.2008.01.006. Epub 2008 Mar 7. PMID 18316142
- [Background] Traber MG, Stevens JF. Vitamins C and E: beneficial effects from a mechanistic perspective. Free Radic Biol Med. 2011 Sep 1;51(5):1000-13. doi: 10.1016/j.freeradbiomed.2011.05.017. Epub 2011 May 25. PMID 21664268
- [Background] Cereda E, Klersy C, Serioli M, Crespi A, D'Andrea F; OligoElement Sore Trial Study Group. A nutritional formula enriched with arginine, zinc, and antioxidants for the healing of pressure ulcers: a randomized trial. Ann Intern Med. 2015 Feb 3;162(3):167-74. doi: 10.7326/M14-0696. PMID 25643304
- [Background] Leigh B, Desneves K, Rafferty J, Pearce L, King S, Woodward MC, Brown D, Martin R, Crowe TC. The effect of different doses of an arginine-containing supplement on the healing of pressure ulcers. J Wound Care. 2012 Mar;21(3):150-6. doi: 10.12968/jowc.2012.21.3.150. PMID 22399084
- [Background] Desneves KJ, Todorovic BE, Cassar A, Crowe TC. Treatment with supplementary arginine, vitamin C and zinc in patients with pressure ulcers: a randomised controlled trial. Clin Nutr. 2005 Dec;24(6):979-87. doi: 10.1016/j.clnu.2005.06.011. Epub 2005 Nov 15. PMID 16297506
- [Background] Theilla M, Schwartz B, Cohen J, Shapiro H, Anbar R, Singer P. Impact of a nutritional formula enriched in fish oil and micronutrients on pressure ulcers in critical care patients. Am J Crit Care. 2012 Jul;21(4):e102-9. doi: 10.4037/ajcc2012187. PMID 22751375
- See also: Incidence of diabetic foot ulcer and lower extremity amputation among Medicare beneficiaries, 2006 to 2008: Data Points #2. — http://www.ncbi.nlm.nih.gov/books/NBK65149/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care Group | Immunonutrition Supplementation Group
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Ineligible patient | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only one study subject enrolled and study was closed one month later. The study subject was enrolled to the no supplement arm; no subjects enrolled to treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Group | Immunonutrition Supplementation Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (0) |  | 63 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Effect of Supplemental Immunonutrition on Wound Healing in Patients With Diabetic Foot Ulcers as Assessed by the Pressure Ulcer Scale for Healing (PUSH) Tool 3.0.
Description: The PUSH Tool 3.0 will be used to score ulcers based on size (cm2), exudate amount, and tissue type present. The score ranges for size, exudate amount, and tissue type are 0-10, 0-3, and 0-4, respectively. For all categories, a higher score indicates a more severe ulcer. The score for each category is combined to generate a final score ranging from 0-17. A higher final score indicates a more severe ulcer. The treating physician will record ulcer scores using this tool at the time of consent and 6 weeks for both the standard of care group and experimental group and calculate the change in ulcer scores from consent to 6 weeks.
Time Frame: 6 weeks
Population: Only one study subject enrolled before study was closed and participant was withdrawn before 6 weeks. The study subject was enrolled to the no supplement arm; no subjects enrolled to treatment arm.
Arm/Group | Standard of Care Group | Immunonutrition Supplementation Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Effect of Supplemental Immunonutrition on Patient Reported Pain Scores in Patients With Diabetic Foot Ulcers.
Description: Patients in both the standard of care and experimental groups will report visual analog scale (VAS) pain scores at 6 weeks.
Time Frame: 6 weeks
Population: as for outcome 1
Arm/Group | Standard of Care Group | Immunonutrition Supplementation Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Effect of Supplemental Immunonutrition on Patient Satisfaction in Patients With Diabetic Foot Ulcers.
Description: Patients in experimental group will complete a survey detailing their satisfaction with the supplemental immunonutrition regimen following completion of study participation. Patients will be asked to rate their satisfaction from very satisfied to very unsatisfied and questions regarding their likelihood to partake in the same treatment regimen for a subsequent ulcer, recommend this treatment regimen to others, and the level of difficulty associated with taking the supplementation.
Time Frame: 6 weeks
Population: as for outcome 1
Arm/Group | Standard of Care Group | Immunonutrition Supplementation Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Long Term Effect of Supplemental Immunonutrition on Wound Healing in Patients With Diabetic Foot Ulcers on Rates of Ulcer Recurrence, Infection, Surgical Intervention, and Amputation.
Description: Study participants in both the standard of care and experimental groups will be monitored via chart review for one year following the completion of their study participation to assess recurrence rates of diabetic foot ulcers and to identify rate of infection, surgical intervention, and amputation.
Time Frame: 1 year
Population: Only one study subject enrolled before study was closed and participant was withdrawn before 1 year. The study subject was enrolled to the no supplement arm; no subjects enrolled to treatment arm.
Arm/Group | Standard of Care Group | Immunonutrition Supplementation Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: Only one study subject enrolled and study was closed one month later. The study subject was enrolled to the no supplement arm; no subjects enrolled to treatment arm.
Arm/Group | Standard of Care Group | Immunonutrition Supplementation Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT05281562/Prot_SAP_001.pdf